CLINICAL TRIAL: NCT02073110
Title: Optical Biopsy to Improve the Diagnosis of Kidney Cancer: a Prospective, Observational, Multicentre, In-vivo Study
Brief Title: Optical Biopsy to Improve the Diagnosis of Kidney Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, P.G.K. Wagstaff, MD., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL41985.018.12
Record Dates: First submitted 2014-02-20; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Cancer
Keywords: Kidney cancer; Renal mass; Small renal mass; Optical Coherence Tomography; OCT; Diffuse Reflectance Spectroscopy; DRS; Optical Biopsy; OB
MeSH Terms: conditions — Kidney Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ≥ 18 years, solid enhancing renal mass suspected for RCC
  Interventions: Device: Percutaneous Optical Biopsy (OCT and DRS)

INTERVENTIONS:
Device: Percutaneous Optical Biopsy (OCT and DRS)

SUMMARY:
Data from the American Cancer Society shows a 70% increase in incidence of kidney and renal pelvis cancer between 2000 and 2010. This increase is attributed to small renal masses (SRM) that are incidentally discovered by abdominal radiological imaging. However, 30% of resected SRMs appear benign on histological examination. Conventional biopsy is currently used to provide pathological information prior to resection. However, its non-diagnostic value is high, up to 33% in SRMs, showing the need for diagnostic improvement.

The investigators have shown that optical biopsy (OB) can differentiate malignant from benign tissue and tumor subtypes. However, translation to the clinic requires a phase 2 clinical study. The investigators will use an OB probe that can be combined with a needle puncture during classical biopsy procedures, additionally providing real time micro-scale images containing quantitative information about tissue properties. The investigators are convinced that OB will greatly improve the diagnosis of renal tumor pathology.

DETAILED DESCRIPTION:
Rationale:

Renal biopsies can be used in patients with renal mass lesions to diagnose whether it concerns a malignant or benign mass. In case of malignancy, surgery will be the following step. However, 7 to 33% of biopsies are non-diagnostic, what can result in unnecessary surgery (even up to 30% in small renal masses). The investigators think that optical biopsy (OB), a new diagnostic tool based on the absorption en reflection of light in tissues, reduces the non-diagnostic biopsy rate. This could have a direct impact on the quality of life of the patients that are therefore scheduled for an unnecessary surgical procedure. Also, concerns about overtreatment have led to the concept of focal therapy, a selective patient tailored nephron sparing surgical or ablation technique of a lesion, reducing lifetime morbidity and side effects without compromising life expectancy. For this novel form of treatment, accurate identification, grading and demarcation of a lesion is crucial and OB is the ideal platform to provide this approach to an improved cure.

Objectives:

Primary

- The accuracy of DRS and OCT in the diagnostic of renal malignancy

Secondary

* The accuracy of DRS and OCT in the diagnostic of renal malignancy and in distinguishing among the 3 main RCC subtypes
* The accuracy of the combination of the DRS and OCT

Study design:

This is a prospective, observational, multi-centre in-vivo study.

Study population:

Patients ≥ 18 years of age, with a solid enhancing renal mass suspected for renal cell carcinoma (RCC) and candidates for active (surgical) treatment of the renal mass.

Intervention:

Patients will receive an ultrasound guided percutaneous OB followed by a Core biopsy (CB) during the same procedure. The planned institutional surgical protocol will be followed irrespective of the results of OB and CB. During surgery (radical/partial, open/laparoscopic, percutaneous ablation) a new set of DRS and OCT measurements of the tumor and normal tissue will be performed.

Main study parameters/endpoints:

1. To determine the accuracy of OB to differentiate renal tumor pathology from benign tissue by means of minimal invasive quantitative DRS and OCT.
2. To determine the differentiation capability of OCT this combined technique to distinguish between the three most common RCC sub-types.
3. To determine whether OB is a good alternative to the percutaneous biopsy for diagnosing renal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Solid, enhancing mass on cross sectional imaging suspect for RCC
* Scheduled for total or partial nephrectomy or for laparoscopic cryoablation.
* Signed informed consent

Exclusion Criteria:

* Patients with a renal mass that are not candidates for active treatment will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age, with a solid enhancing renal mass suspected for renal cell carcinoma (RCC) and candidates for active (surgical) treatment of the renal mass.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of DRS and OCT in the detection of renal malignancy | Participants will undergo OCT/DRS measurements within 2 weeks after inclusion
  By measuring the OCT attenuation coefficient (µOCT) and the DRS optical blood absorption (µaHb), and correlating these values to the histopathology results.

SECONDARY OUTCOMES:
The sensitivity and specificity of DRS and OCT in differentiating between the three main RCC subtypes | Participants will undergo OCT/DRS measurements within 2 weeks after inclusion
  By measuring the OCT attenuation coefficient (µOCT) and the DRS optical blood absorption (µaHb), and correlating these values to the histopathology results.

CONTACTS AND LOCATIONS:
Overall Officials: MP Laguna Pes, MD. PhD., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); JJMCH de la Rosette, MD. PhD., Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Free University Medical Center, Amsterdam
  - Academic Medical Center, Amsterdam

REFERENCES:
- [Derived] Buijs M, Wagstaff PGK, de Bruin DM, Zondervan PJ, Savci-Heijink CD, van Delden OM, van Leeuwen TG, van Moorselaar RJA, de la Rosette JJMCH, Laguna Pes MP. An In-vivo Prospective Study of the Diagnostic Yield and Accuracy of Optical Biopsy Compared with Conventional Renal Mass Biopsy for the Diagnosis of Renal Cell Carcinoma: The Interim Analysis. Eur Urol Focus. 2018 Dec;4(6):978-985. doi: 10.1016/j.euf.2017.10.002. Epub 2017 Oct 24. PMID 29079496